CLINICAL TRIAL: NCT03102918
Title: Cannabidiol Pharmacotherapy for Adults With Cannabis Use Disorder
Acronym: CBD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Kevin P. Hill, MD, MHS, Assistant Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P002013
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Cannabis Use Disorder
Keywords: Cannabidiol
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: In this randomized, double-blind, placebo-controlled trial, cannabis-dependent subjects ages 18-65 will receive medical management over a 6-week period, with half receiving Epidiolex treatment and half receiving placebo.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Active Comparator): Epidiolex
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Participants will receive either up to 800 mg Epidiolex over a 6-week treatment period.
  Other Names: Epidiolex
  Arms: Cannabidiol
Drug: Placebo — Participants will receive placebo over a 6-week treatment period.
  Arms: Placebo

SUMMARY:
Investigators aim to determine Epidiolex's promise as a pharmacotherapy for cannabis use disorder. Investigators hypothesize that Epidiolex, when added to medical management, will result in greater reductions in marijuana use compared to placebo as measured by the 2 primary outcome measures: 1) quantitative THC levels and 2) self-report by Timeline Follow Back. Secondary outcome measures will include treatment retention, patient satisfaction, cannabis withdrawal, cannabis craving, depressive symptoms, anxiety symptoms, , compliance, and cigarette use.

DETAILED DESCRIPTION:
Investigators will conduct a Stage 1 pilot feasibility study at McLean Hospital to begin to evaluate Epidiolex as a pharmacotherapy for adults with cannabis use disorder. In this randomized, double-blind, placebo-controlled trial, cannabis-dependent subjects ages 18-65 will receive medical management over a 6-week period, with half receiving Epidiolex treatment and half receiving placebo. Participants will receive either up to 800 mg Epidiolex or placebo over a 6-week treatment period. Following treatment completion, participants will have a follow-up visits at 10 and 14 weeks. Primary outcomes will include self-report of cannabis smoking and results of quantitative urine drug screens for cannabis. Secondary outcome measures will include treatment retention, patient satisfaction, cannabis withdrawal, cannabis craving, depressive symptoms, anxiety symptoms, compliance, and cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65 years
* DSM 5 diagnosis of cannabis use disorder, based on the Structured Clinical Interview for DSM 5 (SCID-5)
* Express a desire to quit cannabis use within the next 30 days
* Have used cannabis on ≥4 days within the past 30 days (i.e., an average of ≥1 day per week)
* For women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests; for men, contraception will be discussed at the beginning of the study with the study physician
* Consent for us to communicate with their prescribing clinician
* Furnish the names of 2 locators, who would assist study staff in locating them during the study period
* Live close enough to McLean Hospital to attend study visits
* Plan to stay in the Boston area for the next 3 months
* Are willing and able to sign informed consent

Exclusion Criteria:

* Current diagnosis of other drug or alcohol dependence (excluding nicotine)
* Recent (within 3 months) significant cardiac disease
* Current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder
* Current medical condition (including significant laboratory abnormalities, such as abnormal liver function tests) that could prevent regular study attendance
* Mental retardation or organic mental disorder
* Acutely dangerous or suicidal behavior
* Currently in a residential treatment setting in which substance use is monitored and restricted, since the restricted access to drugs could represent an important confounding variable
* Pregnant, nursing, or, if a woman of childbearing potential, not using a form of birth control judged by the investigator to be effective
* Concomitant daily treatment with opioid analgesics, sedative hypnotics, or other known CNS depressants
* Known hypersensitivity to cannabinoids or sesame oil
* Disease of the gastrointestinal system, liver, or kidneys that may impede metabolism or excretion of CBD
* Inability to read or write in English
* History of seizures, head trauma or other history of CNS insult that could predispose the subject to seizures
* Currently taking valproic acid, lamotrigine, or propranolol, medication metabolized by UGT1A9 or UGT2B7 enzymes (CBD may affect these UGT levels)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-20 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol | Placebo
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (10.7) | 28.0 (12.3) | 30.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Self-report Cannabis Use during Baseline [Mean (Standard Deviation); unit: Inhalations per day] — Self-report via Timeline Followback of the number of inhalations per day during the Baseline time period
  Inhalations per day | 26.03 (22.03) | 21.03 (26.61) | 23.53 (23.18)

OUTCOME MEASURES:

1. Primary Outcome: Self-report Instruments to Measure Cannabis Use
Description: Self-reported cannabis inhalations per day during Week 6 as reported by Timeline Followback
Time Frame: During Week 6
Population: One subject in the Cannabidiol arm was withdrawn from the study before Week 6 due to poor medication adherence.
Measure: Mean (Standard Deviation); unit: Inhalations of Cannabis Per Day
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 4 | 5
Inhalations of Cannabis Per Day | 26.72 (26.96) | 5.256 (4.34)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through-out the course of the study during each study visit. This is from baseline until Week 14 when the last follow-up visit was conducted.
Description: Study staff collected any adverse event data during every study visit for each subject. This amounted to twice a week during the study.
Arm/Group | Cannabidiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Due to the small sample size, more subjects would need to be included to be able to draw definitive conclusions from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03102918/Prot_SAP_000.pdf